CLINICAL TRIAL: NCT01676714
Title: Phase II Study of Dovitinib and Pilot Study of Fibroblast Growth Factor Receptor Biomarkers in Advanced Non-Small Cell Lung Cancer or Advanced Colorectal Cancer Previously Treated With Anti-Vascular Endothelial Growth Factor Therapy
Brief Title: Study of Dovitinib and Biomarkers in Advanced Non-Small Cell Lung Cancer or Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#231; 344991 (Other Grant/Funding Number: UC Davis); CTKI258AUS21T (Other Grant/Funding Number: Novartis)
Record Dates: First submitted 2012-08-27; First posted 2012-08-31 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer
Keywords: Dovitinib; Fibroblast Growth Factor Receptor Biomarkers; Anti-Vascular Endothelial Growth Factor Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dovitinib (Experimental): 500 mg of dovitinib (5 capsules) once a day for 5 continuous days and stop for 2 days. Continue to take dovitinib capsules in this manner until until progression or unacceptable toxicity develops.
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib
  Other Names: TK1258

SUMMARY:
The purpose of this study is to find out if dovitinib is an effective treatment for patients with advanced lung cancer or advanced colorectal cancer (CRC) who have progressed on anti-vascular endothelial growth factor (VEGF) treatment.

DETAILED DESCRIPTION:
The purposes of this study are 1) to evaluate the clinical efficacy of dovitinib and 2) to prospectively estimate the prevalence of fibroblast growth factor (FGF) signaling alterations in patients with advanced non-squamous non small cell lung cancer (NSCLC) or advanced CRC who have progressed on anti-VEGF treatment. Additionally, the investigators will make exploratory initial observations of the relationship between FGF signaling alterations and the clinical activity of dovitinib. This trial is expected to provide key biologic information that will inform the clinical development of dovitinib and provide initial evaluation of the analytic characteristics of these potential predictive biomarkers of its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer or colorectal cancer for which no potentially curative treatment options are available
* Any number of prior treatment regimens are allowed
* Immediate prior treatment regimen must have included an anti-VEGF agent. Acceptable anti-VEGF therapy includes bevacizumab, sunitinib, or sorafenib. For other anti-VEGF therapies, contact the principal investigator.
* Last dose administered of bevacizumab must be at least 21-days but not more than 56-days from enrollment.
* Last dose of anti-VEGF tyrosine kinase inhibitor must be at least 7-days but not more than 56-days from enrollment.
* Willingness to consent to research biopsy
* Measurable disease by RECIST 1.1 criteria
* Available tumor site amenable to core needle biopsy as determined by the treating investigator. Any questions regarding suitability of site for biopsy will be adjudicated by the principal investigator.
* Zubrod (ECOG) performance status 0 or 1
* Age ≥ 18 years old
* Patients who give a written informed consent
* Patients must have the following laboratory values:

  * Platelets ≥ 100 x 109/L
  * Absolute neutrophil count ≥ 1.5 x 109/L Hemoglobin > 9 g/dL
  * Serum total bilirubin: ≤ 1.5 x upper limit of normal ULN
  * ALT and AST ≤ 3.0 x ULN ( with or without liver metastases)
  * Serum creatinine ≤ 1.5 x ULN or serum creatinine >1.5 - 3 x ULN

Exclusion Criteria:

* Patients with known brain metastases
* Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer
* Patients who have received the last administration of an anticancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies that have not resolved to NCI CTCAE grade 1 or less.
* Patients who have received the last administration of nitrosurea or mitomycin-C ≤ 6 weeks prior to starting study drug, or who have side effects that have not resolved to NCI CTCAE grade 1 or less.
* Patients who have received targeted therapy ≤ 1 week prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug, or ≤ 2 weeks prior to starting study drug in the case of localized radiotherapy or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery, open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Impaired cardiac function or clinically significant cardiac diseases
  * Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib
  * Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
  * Known diagnosis of human immunodeficiency virus infection
  * Patients who are currently receiving anticoagulation treatment with therapeutic doses of warfarin
  * Other concurrent severe and/or uncontrolled concomitant medical conditions
* Pregnant or breast-feeding women
* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception.
* Fertile males not willing to use contraception, as stated above
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Semrad, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dovitinib
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dovitinib: 500 mg of dovitinib (5 capsules) once a day for 5 continuous days and stop for 2 days. Continue to take dovitinib capsules in this manner until until progression or unacceptable toxicity develops.
  Dovitinib
Arm/Group | Dovitinib
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 100 months
Measure: Count of Participants; unit: Participants
Groups:
- Dovitinib: 500 mg of dovitinib (5 capsules) once a day for 5 continuous days and stop for 2 days.
Arm/Group | Dovitinib
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Disease Control Rate
Description: The total number of patients who demonstrate a response to treatment. Measured by RECIST 1.1 criteria.
Time Frame: From start of treatment, up to 8 weeks
Population: 500 mg of dovitinib (5 capsules) once a day for 5 continuous days and stop for 2 days. Continue to take dovitinib capsules in this manner until progression or unacceptable toxicity develops.
Measure: Number; unit: participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 7
participants | 1

3. Secondary Outcome: Progression Free Survival
Description: The length of time during and after the treatment of the cancer that a patient lives with the disease but it does not get worse. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment until the date of death from any cause, assessed up to 100 months
Measure: Median (Full Range); unit: months
Arm/Group | Dovitinib
Number analyzed (Participants) | 7
months | 1.9 [0.23 to 4.1]

4. Secondary Outcome: Number of Patients Who Experienced Treatment Related Toxicities
Description: Toxicities will be summarized by the type, severity (by NCI CTCAE), time of onset, duration, and outcome. Toxicity will be graded according to the NCI CTCAE version 4.0.
Time Frame: Starting at screening and then at every visit and then up to 30 days after the last dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 30 days after treatment
Arm/Group | Dovitinib
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=10)
Thrombolic Event (Vascular disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=10)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3)
Edema Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (9)
Malaise (General disorders) | 2 (2)
ALT Increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 8 (8)
AST increased (Investigations) | 5 (5)
Blood Bilirubin Increased (Investigations) | 5 (5)
Cholesterol High (Investigations) | 2 (2)
GCT Increased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 4 (4)
Other - LDH Increased (Investigations) | 2 (2)
Weight Loss (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Hypoatremia (Metabolism and nutrition disorders) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4)
General Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes